CLINICAL TRIAL: NCT01233089
Title: Quality of Life and Ease of Fit, Fitting Children With Contact Lenses
Brief Title: Fitting Children With Contact Lenses
Acronym: COPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-368-C-107; P/346/10/C (Other: University of Waterloo)
Record Dates: First submitted 2010-11-01; First posted 2010-11-03 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2011-09

CONDITIONS: Refractive Error
Keywords: Myopia; contact lenses; children
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CARE (Experimental): Investigational single-vision contact lenses worn bilaterally on a daily wear basis and replaced monthly
  Interventions: Device: Lotrafilcon B contact lens, investigational; Device: Contact lens care system (ClearCare)
- AIR OPTIX AQUA (Active Comparator): Commercially available single-vision contact lenses worn bilaterally on a daily wear basis and replaced monthly
  Interventions: Device: Lotrafilcon B contact lens, commercial (AIR OPTIX AQUA); Device: Contact lens care system (ClearCare)
- AIR OPTIX AQUA MULTIFOCAL (Active Comparator): Commercially available multifocal contact lenses worn bilaterally on a daily wear basis and replaced monthly
  Interventions: Device: Lotrafilcon B multifocal contact lens, commercial (AIR OPTIX AQUA MULTIFOCAL); Device: Contact lens care system (ClearCare)

INTERVENTIONS:
Device: Lotrafilcon B contact lens, investigational — Investigational silicone hydrogel, spherical contact lens worn on a daily wear basis and replaced monthly
  Arms: CARE
Device: Lotrafilcon B contact lens, commercial (AIR OPTIX AQUA) — Commercially available silicone hydrogel, spherical contact lens worn on a daily wear basis and replaced monthly.
  Other Names: AIR OPTIX AQUA
  Arms: AIR OPTIX AQUA
Device: Lotrafilcon B multifocal contact lens, commercial (AIR OPTIX AQUA MULTIFOCAL) — Commercially available silicone hydrogel, multifocal, contact lens worn on a daily wear basis and replaced monthly.
  Other Names: AIR OPTIX AQUA MULTIFOCAL
  Arms: AIR OPTIX AQUA MULTIFOCAL
Device: Contact lens care system (ClearCare) — Commercially available, hydrogen peroxide-based system for cleaning, disinfecting, and storing contact lenses
  Other Names: CLEAR CARE

SUMMARY:
The purpose of this three-month study is to compare the quality of life and ease of fit among children wearing investigational single-vision contact lenses, commercially marketed single-vision contact lenses, and commercially marketed multifocal contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Is between 8 and 16 years of age.
* Has the permission of a parent/legal guardian.
* Is willing and able to, or has a parent/legal guardian who is willing and able to help them, follow instructions and maintain the appointment schedule.
* Has had an ocular examination in the last two years.
* Has never worn contact lenses before.
* Has clear corneas and no active ocular disease.
* Can be successfully fit with the lenses to be used in the study.
* Has 20/25 or better best corrected visual acuity in each eye.
* Other protocol-defined inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Has any ocular disease.
* Has a systemic condition that may affect a study outcome variable.
* Is using any systemic or topical medications that may affect ocular health.
* Has ocular or systemic allergies that could interfere with contact lens wear.
* Has any ocular pathology or condition that would affect the wearing of contact lenses.
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 194 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 3 months
Ease of fit | 1 week
  A participant was deemed to be successfully fit if they could insert/remove, handle and maintain study lenses by the 1-week visit and continued in the study.
PREP score | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada

REFERENCES:
- [Result] Paquette L, Jones DA, Sears M, Nandakumar K, Woods CA. Contact lens fitting and training in a child and youth population. Cont Lens Anterior Eye. 2015 Dec;38(6):419-23. doi: 10.1016/j.clae.2015.05.002. Epub 2015 Jun 9. PMID 26070228